CLINICAL TRIAL: NCT03847051
Title: EPIMix (Echo Planar Imaging Mix) Versus CT Brain Pediatric Study
Brief Title: EPIMix Versus CT Brain Pediatric Study
Status: Completed | Type: Observational
Sponsor: Karolinska University Hospital (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Principal Investigator, Anna Falk Delgado, Principal Investigator, Medical doctor, PhD, Specialist in Neuroradiology, Karolinska University Hospital
Other Study IDs: EPIMix pediatric
Record Dates: First submitted 2019-02-12; First posted 2019-02-20 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Brain Diseases
Keywords: MRI (magnetic resonance imaging); Neuroradiology; EPIMix (Echo planar imaging mix); Multicontrast EPI (echo planar imaging); Clinical validation
MeSH Terms: conditions — Brain Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: MRI — Brain MRI without intravenous contrast

SUMMARY:
This study aims to assess the diagnostic feasibility and diagnostic performance of a new fast MR sequence EPIMix for neuroradiological evaluation in comparison to computed tomography of brain in pediatric population.

DETAILED DESCRIPTION:
The study aims to assess the feasibility of fast MR sequence for neuroradiological evaluation in comparison to computed tomography of brain in pediatric population. Imaging quality is analysed with regards to artefacts and lesion conspicuity as well as its diagnostic potential in rendering a probable diagnosis. The primary study aim is to define feasibility and the AUC for diagnostic performance of minute MRI compared to computed tomography.

Included patients are children age 4-18 with suspicion of cerebral pathology with referral to elective computed tomography of the brain.

Study participants are in addition to computed tomography investigated during same day at 3T MR.

ELIGIBILITY:
Inclusion Criteria:

* Age 4-18 years.
* Patient with suspicion of cerebral pathology.
* Referral to elective brain CT study.

Exclusion Criteria:

* CT planned with sedation
* known previous cerebral pathology (follow up study)
* Emergency CT
* Aborted MR exam

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Child with indication for elective brain CT.
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2019-02-15 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Tolerance of a new fast MR method in children | At 0 hours
  Number of aborted MR
Diagnostic potential | At 0 hours
  Diagnostic accuracy to categorize scan as normal or abnormal on a five point Likert scale (1 - definitely normal, 2 - Probably normal, 3 - Indeterminate, 4 - Probably abnormal, 5 - Definitely abnormal) compared to abnormal/normal brain CT.

SECONDARY OUTCOMES:
Lesion classification | At 0 hours
  Classification into disease categories (Neoplastic, Ischemic, Hemorrhagic, Infection, Neuroinflammation, Hydrocephalus, Congenital malformation, Indeterminate)
Lesion location determination | At 0 hours
  Anatomical localization of abnormality (Cerebrum, Cerebellum, Brainstem, Intraventricular, Subarachnoid space including basal cisterns, Intra-orbital, Skull/Skull base/dural, Other)
Diagnostic imaging quality | At 0 hours
  Diagnostic imaging quality (5 point Likert scale; 1 - Excellent diagnostic imaging quality, 2 - Good diagnostic imaging quality, 3 - Sufficient diagnostic imaging quality, 4 - Restricted diagnostic imaging quality, 5 - Poor diagnostic imaging quality)
Lesion description | At 0 hours
  For example effect on brain parenchyma and size
Diagnostic confidence | At 0 hours
  Five point Likert scale (Very confident, Predominantly confident, Fairly confident, Only slightly confident, Not at all confident)
Clinical diagnostic summary report | At 0 hours
  Text (one sentence summary of the finding including type of lesion and location)
Ability to rule out diseases | At 0 hours
  A list of diseases. Number of positive versus negative cases for each investigation (including: Tumor, Abscess, Parenchymal Haemorrhage, Acute Ischemia, Hydrocephalus, Neuroinflammation, Subarachnoid hemorrhage, Extraaxial fluid collection)
Artefacts | At 0 hours
  Artefacts and impact (Motion, Beam hardening, Other) defined as; Not present, Not affecting diagnostic confidence, Degrading diagnostic confidence)

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] De Luca F, Kits A, Martin Munoz D, Aspelin A, Kvist O, Osterman Y, Diaz Ruiz S, Skare S, Falk Delgado A. Elective one-minute full brain multi-contrast MRI versus brain CT in pediatric patients: a prospective feasibility study. BMC Med Imaging. 2024 Jan 24;24(1):23. doi: 10.1186/s12880-024-01196-6. PMID 38267889